CLINICAL TRIAL: NCT02802839
Title: The Use of Virtual Reality in the Reduction of Pain and Anxiety During Venipuncture in Children With Cystic Fibrosis: a Randomized Controlled Trial
Brief Title: Virtual Reality for the Reduction of Pain During Venipuncture in Children With CF
Acronym: VRAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Filippo Festini, Professor of Nursing, University of Florence
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: vers 1 del 15.02.16
Record Dates: First submitted 2016-06-06; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis
Keywords: Virtual Reality; venipuncture
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sperimental (Experimental): The patient will be shown the headset for VR and a selection of age appropriate virtual realities to immerge in by the nurse not performing the procedure. There will be two lists of VRs to choose from, one for age 6 to 12 and one for age 12 to 18 with the following themes: amusement rides /carousel, space rides, zoo, safari, dinosaurs, city touring, landscapes, caverns. Once the patient is ready to wear the headset the application will start and 120 seconds later the procedure will take place. The nurse performing venipuncture will be a different one than the one handling distraction. Once the procedure ends the video will last for one more minute or up to the child' s desire. Only the first venipuncture attempt will be observed.
  Interventions: Device: Virtual Reality
- Observational (No Intervention): Control intervention When arriving to the CF centre for routine visit that implies also the taking of blood samples, after having obtained the informed consent, a trained nurse of the CF Centre, will apply to each child recruited -in the presence of the parent, who may hold the child- the anesthetic cream. Only the first venipuncture attempt will be observed.

INTERVENTIONS:
Device: Virtual Reality
  Arms: Sperimental

SUMMARY:
Children with Cystic fibrosis (CF) have to undergo several needle-related procedures during outpatient visits or hospital stay. It is common for children with CF to display distress and behavioural problems during invasive procedures. Children with chronic diseases have a lower threshold of pain compared to non-chronic patients. Effective management of needle distress in children with CF is critical. Although pharmacological and non pharmacological methods are used during needle -related procedures to lower painful stimuli nearly all patients with CF experience anxiety. Distraction has been shown to be an effective technique that directs children's attention away from noxious stimuli. The application of Virtual Reality (VR) in the medical field has been shown to be successful already 15 years ago. VR has found its use during the medication of burns and in patients undergoing cancer treatments whereas so far few studies have been published to assess its efficacy in reducing needle related pain and distress in children and none in children with CF.

Objectives To assess the efficacy of VR in reducing pain and distress during venipuncture in children with CF compared to routine care.

Project description Randomized controlled parallel trial with a 1 to 1 allocation ratio. The use of VR compared to standard care during venipuncture in children with CF (age 6-18 years) attending the outpatient clinic of the CF Centre of Florence will be compared over the period of 1 year. Patients randomly assigned to arm A will use VR during the procedure, those patients assigned to arm B will receive routine care.

Anticipated output Determination of the efficacy of VR in lowering pain and distress during venipuncture.

DETAILED DESCRIPTION:
Research Plan: Background, Specific Aims and Rationale Background Cystic fibrosis (CF), the most common lethal genetic disorder in Caucasians, affects over 80,000 patients worldwide. Its incidence is calculated as occurring in one out of every 2,500 living newborns. Advances in the care of CF patients have been associated with impressive increases in survival during the last 30 years. The mean life expectancy for patients now diagnosed by newborn screening approaches 40 years and approximately 47% of Italian patients are 18 years of age or older. This striking result is mainly due to better treatment of bacterial lung infections, the main cause of pulmonary deterioration and early death of the patients. To be efficacious early diagnose and treatment are of fundamental importance this is why patients are routinely visited and tested several times during the year. Tests include also the collection of blood samples to detect and monitor infections and general health conditions. This means that after the diagnose of CF, children undergo at least 1 blood sample per year among other sample collections as sputum or throat swabs. Antibiotic intravenous treatment is not uncommon in these patients and involves the positioning of peripheral venous catheters (pvc), midlines or central venous access. As shown in previous studies it is common for children with CF to display distress and behavioural problems during invasive procedures. Like other children with chronic diseases children with CF have a lower threshold of pain compared to non-chronic patients as shown by data published by this research group. In fact there is a common belief among nurses and healthcare professionals that children, subject to repeated procedures, feel less pain because of a higher pain threshold compared to children who only sporadically visit the hospital. This misconception may lead professionals to lower their attention for the prevention and treatment of pain in children with chronic diseases. The purpose of the study of Bisogni was to compare the pain perceived and the behavioural distress shown during a standardized venipuncture by children with chronic diseases who have already been exposed to venipuncture, with those of a group of children who have never had any previous experience of venipuncture before. The results show that chronic children reported a median pain score of 8 on the Wong numeric scale, while non-chronic children reported a median pain score of 2. The results were statistically significant indicating that children subject to continue venipuncture procedures have a lower pain threshold than children of the same sex and age who experience venipuncture for the first time. This findings show that in daily clinical practice it is always necessary to promote effective and validated techniques to support patients for the reduction of pain and distress especially in chronic children who will need lifelong treatments and where anticipatory distress is very common. In fact nearly all patients with CF experience anticipatory pain. Anticipatory anxiety may be explained as a condition which precedes an event or an action where one thinks of the painful experience even before the actual painful stimuli occur. This leads children to live with high concern and fear the periodic hospital visits leading them to react in fight, flight or freeze mode and with their acute stress response affecting also parents and nurses behaviour. Different pharmacological and non pharmacological methods are already widely used during needle related procedures to try to lower pain and distress.

Specific Aims and Rationale The primary aim of this study is to assess the efficacy of VR as a distraction technique during the procedure of venipuncture for blood tests in children with CF in regards to anticipatory distress and pain. The parent ratings of their child's fear and pain and the nurse ratings of children's distress and cooperation will also be assessed.

Distraction has been shown to be an effective non pharmacological technique and is often defined as a strategy-whether cognitive or behavioral- that draws a child's attention away from noxious pain stimuli. Kleiber and Harper draw further distinctions and define distraction as a cognitive coping strategy that passively redirects the subject's attention or actively involves the subject with a task. Despite its widespread use, "there is no universally accepted theory to explain the function of distraction".

VR puts the patient in a different dimension allowing him to immerge into a different dimension shutting out what is going on around him. Patients will be able to choose among an age appropriate choice of VR apps. VR is believed to hold an advantage over other distraction techniques by virtue of its cocoon-like equipment and its engaging and immersive nature. Set in an enclosed headset, VR provides the opportunity for a mental escape by strategically drawing individuals into an alternative world. By controlling their perceptual environment, patients can redirect multiple senses from a hospital environment to one involving positive and entertaining activities.

The application of VR in the medical field has been shown to be successful already 15 years ago. VR has found its use during the medication of burns and in patients undergoing cancer treatments whereas so far few studies have been published to assess its efficacy in reducing needle related pain and distress in children and none in children with CF.

Koller in her review concludes that VR is a complex and costly method that holds promise as an effective intervention. However today the costs of such devices are more affordable starting from 6 euro for a cardboard device and up to 80 Euro for more sophisticated headsets, making this technique easily implemented. Several authors have called for larger sample sizes and more heterogeneous participants to determine how VR can be used most effectively.

ELIGIBILITY:
Inclusion Criteria:

* CF diagnosed by at least two sweat test according to Gibson and Cook (Legrys 1996)
* age from 6 to 18
* regularly attending the CF centre of Florence
* who do not wear glasses, do not have amblyopia, who do not have monocular vision
* who have not taken pain medications in the last 8 hours
* child's and parent's assent of the informed consent

Exclusion Criteria:

* CF not diagnosed not diagnosed according to Gibson and Cook
* under the age of 6 years and over the age of 18
* not regularly attending the CF centre of Florence
* who wear glasses, who have amblyopia, who have a monocular vision
* who have taken pain medications in the last 8 hours
* child's or parent's dissent of the informed consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pain | 30 seconds after the procedure
  Vas-Pain scale self administered by the patient and the parent

SECONDARY OUTCOMES:
Anxiety | before the procedure
  Anxiety VAS consists of a 10-cm horizontal line, anchored on the left by the words ''not at all anxious'' and on the right by ''extremely anxious.'' A higher score indicates greater anxiety (Daveya 2007).
Distress | during the procedure
  The m-YPAS Scale is an observational scale that includes five categories of child behavior, giving them a score based on the descriptions provided in the same scale. These behaviors are: Activity (score 1 to 4), Vocalizations (score 1 to 6), Emotional Expressivity (score 1 to 4), State of Apparent Arousal (score 1 to 4), Use of Parents (score 1 to 4). The overall score is calculated by weighing the scores: the score of each category is divided by the number of items in the category. Then, the 5 calculated values in each category are added together and the sum is multiplied by 100 and divided by 5.

OTHER OUTCOMES:
Distress | during the procedure
  Observation Scale of Behavioural Distress Revised (OSBD-R) described by Eliott et al.
Distress | 30 seconds after the procedure
  To measure distress of the patient the nurse performing venipuncture will be asked after the procedure to use a VAS to rate the patient's degree of observed distress during the just completed procedure. The end-points of the 10 centimetre scale for distress are labelled "Not Distressed" and "Very Distressed" (Powers et al., 1993).
Cooperation | 30 seconds after the procedure
  To measure cooperation of the patient the nurse performing venipuncture will be asked after the procedure to use a VAS to rate the patient's degree of cooperation during the just completed procedure. The end-points of the 10 centimetre scale for cooperation distress are labelled "Not Cooperative" and "Very Cooperative" (Powers et al., 1993).

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Festini, Prof of Nurs, Study Director — Univisersity of Florence
Locations (1):
- Meyer Children Hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duff AJ. Psychological interventions in cystic fibrosis and asthma. Paediatr Respir Rev. 2001 Dec;2(4):350-7. doi: 10.1053/prrv.2001.0171. PMID 12052307
- [Result] Bisogni S, Dini C, Olivini N, Ciofi D, Giusti F, Caprilli S, Gonzalez Lopez JR, Festini F. Perception of venipuncture pain in children suffering from chronic diseases. BMC Res Notes. 2014 Oct 18;7:735. doi: 10.1186/1756-0500-7-735. PMID 25326685
- [Result] Ayers S, Muller I, Mahoney L, Seddon P. Understanding needle-related distress in children with cystic fibrosis. Br J Health Psychol. 2011 May;16(Pt 2):329-43. doi: 10.1348/135910710X506895. Epub 2011 Mar 9. PMID 21489060
- [Result] Sermet-Gaudelus I, De Villartay P, de Dreuzy P, Clairicia M, Vrielynck S, Canoui P, Kirszenbaum M, Singh-Mali I, Agrario L, Salort M, Charron B, Dusser D, Lenoir G, Hubert D. Pain in children and adults with cystic fibrosis: a comparative study. J Pain Symptom Manage. 2009 Aug;38(2):281-90. doi: 10.1016/j.jpainsymman.2008.08.009. Epub 2009 Apr 11. PMID 19364632
- [Result] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481